CLINICAL TRIAL: NCT00487240
Title: Comparison of Two Basal Insulin Analogs (Insulin Lispro Protamine Suspension and Insulin Detemir) in Basal-Bolus Therapy for Patients With Type 1 Diabetes
Brief Title: Comparison of Two Basal Insulin Therapies for Patients With Type 1 Diabetes
Acronym: IOOZ
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Office, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10937; F3Z-MC-IOOZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Results first posted 2009-09-25 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2010-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes; type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin Lispro Protamine Suspension (Experimental): Insulin Lispro Protamine Suspension twice daily
  Interventions: Drug: Insulin Lispro Protamine Suspension
- Detemir (Active Comparator): Insulin Levemir (detemir) subcutaneous (SC) twice daily.
  Interventions: Drug: Insulin Levemir

INTERVENTIONS:
Drug: Insulin Lispro Protamine Suspension — Patient specific dose, twice daily (BID), within 15 minutes before meals, subcutaneous (SC) injection x 32 weeks.
  Other Names: ILPS; NPL; Humalog; LY275585
  Arms: Insulin Lispro Protamine Suspension
Drug: Insulin Levemir — Patient specific dose insulin Levemir (detemir) twice daily (BID) subcutaneous (SC) injection x 32 weeks
  Arms: Detemir

SUMMARY:
The purpose of this study is to examine the efficacy and safety of insulin lispro protamine suspension (ILPS) as compared to insulin detemir as basal insulin combined with mealtime insulin therapy in patients with type 1 diabetes. A gatekeeper strategy will be employed for sequentially testing the secondary objectives.

DETAILED DESCRIPTION:
Phase 3b, randomized, multicenter, multinational, open-label, two-arm, active control, parallel study to determine safety, efficacy, and noninferiority of basal analog insulin lispro protamine suspension (ILPS, also referred to as NPL [neutral protamine Hagedorn]), injected two times a day, compared with basal analog insulin detemir, injected two times a day, as measured by change in hemoglobin A1c (HbA1c) from baseline (Visit 2) to 32 weeks in adult patients with type 1 diabetes when used in combination with bolus insulin lispro, injected three times a day.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes for one year or more
* Age 18 years or older
* Body mass index (BMI) less than or equal to 35 kilograms per square meter (kg/m2)
* Have a hemoglobin A1c (HbA1c) 1.2 to 2.0 times the upper limit of the normal (ULN) reference range within 30 days prior to Visit 1 or collected and analyzed at a local laboratory at Visit 1
* As determined by the investigator, are capable and willing to do the following:

  * perform self monitoring of blood glucose (SMBG),
  * complete patient diaries as required for this protocol,
  * use the insulin injection device(s) according to the instructions provided,
  * are receptive to diabetes education,
  * comply with the required study visits.

Exclusion Criteria:

* Have taken any oral antihyperglycemic medications (OAMs) within 3 months prior to Visit 1.
* Have had more than one episode of severe hypoglycemia, as defined in the Abbreviations and Definitions section of the protocol, within 6 months prior to entry into the study
* Are pregnant or intend to become pregnant during the course of the study or are sexually active women of childbearing potential not actively practicing birth control by a method determined by the investigator to be medically acceptable or women who are breastfeeding
* Are receiving chronic (lasting longer than 14 consecutive days) systemic glucocorticoid therapy (excluding topical, intra-articular, intraocular, and inhaled preparations) or have received such therapy within the 4 weeks immediately preceding Visit 1.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (28):
- United States (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Springfield, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
- Argentina (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Plata
- Australia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wollongong, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fortaleza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Hungary (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mosonmagyaróvár
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pécs
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szentes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zalaegerszeg
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pachuca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Puebla City
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baia Mare
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brasov
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
- Russia (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arkhangelsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rostov-on-Don
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg

REFERENCES:
- [Result] Chacra AR, Kipnes M, Ilag LL, Sarwat S, Giaconia J, Chan J; COMPLETE T1D investigators. Comparison of insulin lispro protamine suspension and insulin detemir in basal-bolus therapy in patients with Type 1 diabetes. Diabet Med. 2010 May;27(5):563-9. doi: 10.1111/j.1464-5491.2010.02986.x. PMID 20536953
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: First 4 weeks (Titration Period): acclimate patients to insulin regimen and optimize insulin dose. Final 28 weeks (Maintenance Period): Minimum of 6 months' stable insulin dosage. 456 patients were screened; 69 did not meet entry criteria and 387 were randomized; 6 patients were excluded from the 387 randomized to create the Full Analysis Set.
Groups:
- Insulin Lispro Protamine Suspension: Patient specific dose insulin lispro protamine suspension, twice daily (BID), within 15 minutes before meals, subcutaneous (SC) injection x 32 weeks
- Detemir: Patient specific dose insulin Levemir (detemir) twice daily (BID) subcutaneous (SC) injection x 32 weeks
Period: Overall Study
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Started | 195 | 192
Full Analysis Set (ITT Population) | 192 | 189
Completed | 164 | 166
Not Completed | 31 | 26
Not completed — Withdrawal by Subject | 12 | 6
Not completed — Lost to Follow-up | 7 | 6
Not completed — Adverse Event | 0 | 4
Not completed — Protocol Violation | 5 | 5
Not completed — Entry Criteria Not Met | 3 | 4
Not completed — Sponsor Decision | 2 | 1
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Lispro Protamine Suspension | Detemir | Total
Number analyzed (Participants) | 192 | 189 | 381
Age Continuous [Mean (Standard Deviation); unit: years] | 36.10 (13.33) | 36.19 (13.09) | 36.14 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 91 | 187
  Male | 96 | 98 | 194
Region of Enrollment [Number; unit: participants]
  United States | 34 | 35 | 69
  Hungary | 16 | 17 | 33
  Mexico | 14 | 12 | 26
  Greece | 16 | 16 | 32
  Argentina | 16 | 16 | 32
  Brazil | 20 | 19 | 39
  Romania | 22 | 21 | 43
  Australia | 17 | 17 | 34
  Russian Federation | 37 | 36 | 73
Race/Ethnicity [Number; unit: participants]
  African | 2 | 1 | 3
  Caucasian | 165 | 160 | 325
  East Asian | 0 | 0 | 0
  Hispanic | 25 | 28 | 53
  Native American | 0 | 0 | 0
  West Asian | 0 | 0 | 0
  Aboriginal and/or Torres Strait Islander | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by square height.
  kilograms per square meter (kg/m^2) | 25.15 (4.17) | 25.46 (4.17) | 25.30 (4.17)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 14.58 (10.69) | 13.83 (9.80) | 14.20 (10.26)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percent of HbA1c] | 8.87 (1.29) | 8.64 (1.27) | 8.75 (1.28)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (HbA1c) From Baseline to Endpoint
Time Frame: baseline and 32 weeks
Population: Number of randomized patients with baseline and at least one post-baseline value. Intent to treat population. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: percent of HbA1c
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 187 | 185
percent of HbA1c
  Baseline | 8.88 (0.10) | 8.68 (0.10)
  Change from Baseline | -0.69 (0.07) | -0.59 (0.07)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Hypothesis: basal analog insulin lispro protamine suspension (ILPS), is inferior to basal analog insulin detemir, as measured by change in HbA1c from baseline to endpoint; Test type: Non-Inferiority or Equivalence — Noninferiority limit of 0.4% using the upper limit of a two-sided test at a significance level of 0.05 with 90% power assuming a 1.1 Standard Deviations (SD); p = 0.332, ANCOVA; ANCOVA Model: Variable=Treatment + Baseline + Country; Mean Difference (Net) = -0.10, 95% CI [-0.29 to 0.10] — Least Squares Mean Difference = Insulin Lispro Protamine Suspension minus Detemir

2. Secondary Outcome: Actual and Change From Baseline Hemoglobin A1c (HbA1c) Values
Description: The summary statistics represents the mean of all subjects. Change from baseline is calculated for each individual subject for the specific visit and then the "mean change from baseline" is calculated by averaging out for all subjects. [Sum over all (i) {A1c at Week 8 for Subject(i) minus A1c Baseline for Subject (i)}/Total Subjects]. Therefore, for example, the Change from Baseline is not equal to the difference of Mean A1c for Week 8 minus Mean A1c for baseline.
Time Frame: Baseline, 8,16, 24, 32 Weeks
Population: Number of randomized patients with baseline and at least one post-baseline value. Intent to treat population.
Measure: Least Squares Mean (Standard Error); unit: percent of HbA1c
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 187 | 185
percent of HbA1c
  Baseline | 8.88 (0.10) | 8.68 (0.10)
  8 Week HbA1c (n=184, n=179) | 8.08 (0.07) | 8.11 (0.07)
  8 Week Change from Baseline | -0.68 (0.07) | -0.64 (0.07)
  16 Week HbA1c (n=174, n=173) | 7.94 (0.07) | 8.08 (0.08)
  16 Week Change from Baseline | -0.81 (0.07) | -0.67 (0.08)
  24 Week HbA1c (n=171, n=174) | 8.07 (0.08) | 8.11 (0.08)
  24 Week Change from Baseline | -0.69 (0.08) | -0.65 (0.08)
  32 Week HbA1c (n=165, n=165) | 8.09 (0.08) | 8.14 (0.08)
  32 Week Change from Baseline | -0.68 (0.08) | -0.62 (0.08)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.718, ANCOVA — P-value for 8 Week Change from Baseline; ANCOVA Model: Variable=Treatment+Baseline+Country; Mean Difference (Net) = -0.03, 95% CI [-0.22 to 0.15] — Least Squares Mean Difference=Insulin Lispro Protamine Suspension minus Detemir
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.187, ANCOVA — P-value for 16 Week Change from Baseline; ANCOVA Model: Variable=Treatment+Baseline+Country; Mean Difference (Net) = -0.14, 95% CI [-0.34 to 0.07] — Least Squares Mean Difference = Insulin Lispro Protamine Suspension minus Detemir
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.704, ANCOVA — P-value for 24 Week Change from Baseline; ANCOVA Model: Variable=Treatment+Baseline+Country; Mean Difference (Net) = -0.04, 95% CI [-0.25 to 0.17] — Least Squares Mean Difference = Insulin Lispro Protamine Suspension minus Detemir
Statistical Analysis 4: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.599, ANCOVA — P-value for 32 Week Change from Baseline; ANCOVA Model: Variable=Treatment+Baseline+Country; Mean Difference (Net) = -0.06, 95% CI [-0.27 to 0.15] — Least Squares Mean Difference = Insulin Lispro Protamine Suspension minus Detemir

3. Secondary Outcome: Percentage of Patients With Hemoglobin A1c (HbA1c) Less Than or Equal to 7.0% and HbA1c Less Than or Equal to 6.5%
Time Frame: 32 Weeks
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 187 | 185
percentage of participants
  With HbA1c ≤7.0% | 18.5 | 18.7
  With HbA1c >7.0% | 81.5 | 81.3
  With HbA1c <7.0% | 15.2 | 15.4
  With HbA1c ≥7.0% | 84.8 | 84.6
  With HbA1c ≤6.5% | 8.7 | 9.9
  With HbA1c >6.5% | 91.3 | 90.1
  With HbA1c <6.5% | 7.1 | 8.2
  With HbA1c ≥6.5% | 92.9 | 91.8
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value for With HbA1c ≤7.0%
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 1.000, Fisher Exact — P-value for With HbA1c <7.0%
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.722, Fisher Exact — P-value for With HbA1c ≤6.5%
Statistical Analysis 4: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.699, Fisher Exact — P-value for With HbA1c <6.5%

4. Secondary Outcome: 7-Point Self-Monitored Blood Glucose (SMBG) at Endpoint
Description: Actual daily mean blood glucose levels at endpoint. The SMBG excursion is the difference between the postprandial and preprandial blood glucose concentration taken at the morning, midday and evening meals.
Time Frame: 32 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 192 | 189
millimoles per Liter (mmol/L)
  Daily Mean 7-Point SMBG (N=164,N=172) | 8.67 (1.97) | 8.48 (1.80)
  Daily Mean Pre-Meal (N=174,N=181) | 8.77 (2.37) | 8.56 (2.10)
  Daily Mean Postprandial Meal (N=168,N=176) | 8.70 (2.08) | 8.58 (2.09)
  Daily Mean Morning+Evening Pre-Meal (N=174,N=181) | 9.00 (2.55) | 8.75 (2.48)
  Actual Morning Pre-Meal (N=175,N=182) | 9.09 (3.18) | 8.62 (3.00)
  Actual Morning Postprandial Meal (N=171,N=178) | 8.68 (2.89) | 8.56 (2.73)
  Actual Midday Pre-Meal (N=175,N=181) | 8.29 (2.92) | 8.19 (2.39)
  Actual Midday Postprandial Meal (N=170,N=177) | 8.54 (2.49) | 8.61 (2.44)
  Actual Evening Pre-Meal (N=174,N=181) | 8.92 (2.72) | 8.87 (2.90)
  Actual Evening Postprandial Meal (N=172,N=181) | 9.05 (2.97) | 8.60 (2.71)
  Actual 0300 Hours (N=167,N=173) | 8.49 (2.85) | 8.29 (2.57)
  Actual Morning SMBG Excursion (N=171,N=178) | -0.34 (2.94) | -0.12 (2.83)
  Actual Midday SMBG Excursion (N=170,N=176) | 0.38 (2.52) | 0.46 (2.59)
  Actual Evening SMBG Excursion (N=172,N=181) | 0.12 (2.72) | -0.24 (3.05)
  Actual Daily Mean SMBG Excursion (N=168,N=176) | 0.06 (1.68) | 0.01 (1.71)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.259, ANCOVA — P-value for Daily Mean 7-Point SMBG; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.468, ANCOVA — P-value for Daily Mean Pre-Meal; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.395, ANCOVA — P-value for Daily Mean Postprandial Meal; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 4: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.414, ANCOVA — P-value for Daily Mean Morning and Evening Pre-Meal; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 5: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.275, ANCOVA — P-value for Actual Morning Pre-Meal; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 6: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.611, ANCOVA — P-value for Actual Morning Postprandial Meal; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 7: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.763, ANCOVA — P-value for Actual Midday Pre-Meal; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 8: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.977, ANCOVA — P-value for Actual Midday Postprandial Meal; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 9: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.586, ANCOVA — P-value for Actual Evening Pre-Meal; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 10: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.093, ANCOVA — P-value for Actual Evening Postprandial Meal; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 11: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.516, ANCOVA — P-value for Actual 0300 Hours; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 12: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.576, ANCOVA — P-value for Actual Morning SMBG Excursion; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 13: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.876, ANCOVA — P-value for Midday SMBG Excursion; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 14: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.261, ANCOVA — P-value for Evening SMBG Excursion; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 15: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.567, ANCOVA — P-value for Daily Mean SMBG Excursion; ANCOVA Model: Variable=Treatment+Baseline+Country

5. Secondary Outcome: Glycemic Variability at Endpoint
Description: Glycemic variability was measured by standard deviation (SD) value of fasting blood glucose as measured by intra-patient glycemic variability (determined by the 7-point self-monitored blood glucose [SMBG] profiles at endpoint); mean value (M-value), which was the mean of the intra-days self-monitored blood glucose values, and by the mean of daily difference (MODD), which was the mean of the between-days self-monitored blood glucose values.
Time Frame: 32 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 187 | 185
millimoles per Liter (mmol/L)
  Standard Deviation (SD) Value (N=172, N=180) | 2.64 (2.09) | 2.30 (1.84)
  Mean Value (M-Value) (N=175, N=182) | 36.39 (31.82) | 32.19 (25.79)
  Mean Daily Difference (MODD) Value (N=172, N=180) | 3.04 (1.90) | 2.78 (1.79)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; If the primary analysis achieves statistical significance at a 0.05 level (that is, the null hypothesis for the primary analysis [primary outcome measure] is rejected), then the first secondary hypothesis (glycemic variability) is tested at an error rate of 0.05; Test type: Non-Inferiority or Equivalence — A noninferiority margin of 0.8 mmol/L was chosen to prove noninferiority of ILPS to detemir; Mean Difference (Net) = 0.36, 95% CI [-0.03 to 0.75] — Least Squares Mean difference = Insulin Lispro Protamine Suspension - Detemir
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.132, ANCOVA — P-value for M-Value; ANCOVA Model: Variable=Treatment+Baseline+Country
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.179, ANCOVA — P-value for MODD; ANCOVA Model: Variable=Treatment+Baseline+Country

6. Secondary Outcome: Number of Self-Reported Hypoglycemic Episodes (Including Nocturnal, Non-Nocturnal, and Severe Hypoglycemia) Overall and at Endpoint
Description: Nocturnal: Defined as any hypoglycemic event that occurs between bedtime and waking. Non-Nocturnal: Defined as any hypoglycemic event that occurs between waking and bedtime. Severe: An episode with symptoms consistent with neuroglycopenia in which the patient requires the assistance of another person; associated with either a blood glucose level of <2.8 mmol/L (<50 mg/dL) or prompt recovery after oral carbohydrate, glucagon, or intravenous glucose.
Time Frame: Baseline to 32 Weeks
Population: as for outcome 1
Measure: Number; unit: episodes of hypoglycemia
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 192 | 189
episodes of hypoglycemia
  Endpoint Hypoglycemic Episodes | 134 | 135
  Overall Hypoglycemic Episodes | 173 | 173
  Endpoint Nocturnal Hypoglycemic Episodes | 69 | 55
  Overall Nocturnal Episodes (N=191,N=186) | 125 | 111
  Endpoint Non-Nocturnal Hypoglycemic Episodes | 127 | 129
  Overall Non-Nocturnal Hypoglycemic Episodes | 172 | 172
  Endpoint Severe Hypoglycemic Episodes | 11 | 3
  Overall Severe Hypoglycemic Episodes (N=171,N=170) | 24 | 13
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.737, Fisher Exact — P-value for Endpoint Hypoglycemic Episodes
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.724, Fisher Exact — P-value for Overall Hypoglycemic Episodes
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.157, Fisher Exact — P-value for Endpoint Nocturnal Hypoglycemic Episodes
Statistical Analysis 4: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.287, Fisher Exact — P-value for Overall Nocturnal Episodes
Statistical Analysis 5: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.664, Fisher Exact — P-value for Endpoint Non-Nocturnal Hypoglycemic Episodes
Statistical Analysis 6: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.730, Fisher Exact — P-value for Overall Non-Nocturnal Hypoglycemic Episodes
Statistical Analysis 7: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.053, Fisher Exact — P-value for Endpoint Severe Hypoglycemic Episodes
Statistical Analysis 8: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.081, Fisher Exact — P-value for Overall Severe Hypoglycemic Episodes

7. Secondary Outcome: 1-Year Adjusted Rates of Self-Reported Hypoglycemic Episodes (Including Nocturnal, Non-Nocturnal, and Severe) Overall and at Endpoint
Description: as for outcome 6
Time Frame: baseline to 32 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hypoglycemic events per 1 year
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 192 | 189
hypoglycemic events per 1 year
  Endpoint Hypoglycemic Rate | 66.41 (90.91) | 52.60 (70.62)
  Overall Hypoglycemic Rate | 76.45 (85.07) | 61.21 (64.25)
  Endpoint Nocturnal Hypoglcemic Rate | 8.90 (18.65) | 5.60 (13.20)
  Overall Nocturnal Hypoglycemic Rate | 9.65 (15.01) | 6.01 (10.31)
  Endpoint Non-Nocturnal Hypoglycemic Rate | 57.08 (83.17) | 46.88 (65.28)
  Overall Non-Nocturnal Hypoglycemic Rate | 66.58 (78.63) | 54.83 (58.94)
  Endpoint Severe Hypoglycemic Rate | 0.63 (3.08) | 0.10 (0.79)
  Overall Severe Hypoglycemic Rate | 0.42 (1.43) | 0.25 (1.26)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.280, ANCOVA — P-value for Endpoint Hypoglycemic Rate; ANCOVA Model: Variable=Treatment+Baseline+Country. Hypoglycemic Rate (Adjusted for 1 year) was used in the analysis
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.193, ANCOVA — P-value for Overall Hypoglycemic Rate; ANCOVA Model: Variable=Treatment+Baseline+Country. Hypoglycemic Rate (Adjusted for 1 year) was used in the analysis
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.042, ANCOVA — P-value for Endpoint Nocturnal Hypoglycemic Rate; ANCOVA Model: Variable=Treatment+Baseline+Country. Hypoglycemic Rate (Adjusted for 1 year) was used in the analysis
Statistical Analysis 4: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value for Overall Nocturnal Hypoglycemic Rate; ANCOVA Model: Variable=Treatment+Baseline+Country. Hypoglycemic Rate (Adjusted for 1 year) was used in the analysis
Statistical Analysis 5: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.579, ANCOVA — P-value for Endpoint Non-Nocturnal Hypoglycemic Rate; ANCOVA Model: Variable=Treatment+Baseline+Country. Hypoglycemic Rate (Adjusted for 1 year) was used in the analysis
Statistical Analysis 6: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.531, ANCOVA — P-value for Overall Non-Nocturnal Hypoglycemic Rate; ANCOVA Model: Variable=Treatment+Baseline+Country. Hypoglycemic Rate (Adjusted for 1 year) was used in the analysis
Statistical Analysis 7: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.017, ANCOVA — P-value for Endpoint Severe Hypoglycemic Rate; ANCOVA Model: Variable=Treatment+Baseline+Country. Hypoglycemic Rate (Adjusted for 1 year) was used in the analysis
Statistical Analysis 8: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.038, ANCOVA — P-value for Overall Severe Hypoglycemic Rate; ANCOVA Model: Variable=Treatment+Baseline+Country. Hypoglycemic Rate (Adjusted for 1 year) was used in the analysis

8. Secondary Outcome: 30-Day Adjusted Rates of Self-Reported Hypoglycemic Episodes (Including Nocturnal, Non-Nocturnal, and Severe) Overall and at Endpoint
Time Frame: baseline to 32 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hypoglycemic events per 30 days
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 192 | 189
hypoglycemic events per 30 days
  Endpoint Hypogylcemic Rate | 5.45 (7.47) | 4.32 (5.80)
  Overall Hypoglycemic Rate | 6.28 (6.99) | 5.03 (5.28)
  Endpoint Nocturnal Hypoglycemic Rate | 0.73 (1.53) | 0.46 (1.08)
  Overall Nocturnal Hypoglycemic Rate | 0.79 (1.23) | 0.49 (0.85)
  Endpoint Non-Nocturnal Hypoglycemic Rate | 4.69 (6.83) | 3.85 (5.36)
  Overall Non-Nocturnal Hypoglycemic Rate | 5.47 (6.46) | 4.50 (4.84)
  Endpoint Severe Hypoglycemic Rate | 0.05 (0.25) | 0.01 (0.06)
  Overall Severe Hypoglycemic Rate | 0.03 (0.12) | 0.02 (0.10)

9. Secondary Outcome: Change From Baseline in Absolute Body Weight at 32 Week Endpoint
Time Frame: Baseline, 32 Weeks
Population: Number of randomized patients with baseline and at least one post-baseline value. Intent to treat population.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 192 | 189
kilograms
  Baseline | 72.76 (15.53) | 72.69 (14.59)
  Change from Baseline | 1.54 (3.18) | 0.58 (3.19)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; If the first secondary null hypothesis (glycemic variability) is rejected, then the second secondary hypothesis (weight change) is tested at an error rate of 0.05; Test type: Non-Inferiority or Equivalence — A noninferiority margin of 1.5 kg was chosen to prove noninferiority of ILPS to detemir; p = 0.003, ANCOVA — P-value for Change from Baseline; ANCOVA Model: Variable=Treatment+Baseline+Country; Mean Difference (Net) = 0.97, 95% CI [0.34 to 1.60] — Least Squares Mean Difference = Insulin Lispro Protamine Suspension minus Detemir

10. Secondary Outcome: Insulin Dose Per Body Weight (Total and By Component [Basal and Bolus])
Description: Total daily insulin dose adjusted for body weight (U/kg/day) was assessed.
Time Frame: 32 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units of insulin per kilogram per day
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 192 | 189
units of insulin per kilogram per day
  Total Insulin (N=192, N=188) | 0.91 (0.30) | 0.99 (0.41)
  Total Bolus Insulin (N=191, N=187) | 0.39 (0.17) | 0.45 (0.22)
  Total Basal Insulin (N=192, N=188) | 0.53 (0.20) | 0.55 (0.26)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.023, ANOVA — P-value for Total Insulin; ANOVA Model: Variable=Treatment+Country
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.004, ANOVA — P-value for Total Bolus Insulin; ANOVA Model: Variable=Treatment+Country
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.282, ANOVA — P-value for Total Basal Insulin; ANOVA Model: Variable=Treatment+Country

11. Secondary Outcome: Insulin Dose (Total and By Component [Basal and Bolus])
Description: Total daily insulin dose (U/day) was assessed.
Time Frame: 32 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units of insulin per day (U/day)
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Number analyzed (Participants) | 192 | 189
units of insulin per day (U/day)
  Total Insulin (N=192, N=188) | 67.78 (27.42) | 73.84 (38.38)
  Total Bolus Insulin (N=191, N=187) | 28.94 (14.69) | 33.32 (20.41)
  Total Basal Insulin (N=192, N=188) | 38.99 (17.37) | 40.70 (22.29)
Statistical Analysis 1: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.82, ANOVA — P-value for Total Insulin; ANOVA Model: Variable=Treatment+Country
Statistical Analysis 2: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.19, ANOVA — P-value for Total Bolus Insulin; ANOVA Model: Variable=Treatment+Country
Statistical Analysis 3: Comparison: Insulin Lispro Protamine Suspension vs Detemir; Test type: Superiority or Other; p = 0.416, ANOVA — P-value for Total Basal Insulin; ANOVA Model: Variable=Treatment+Country

ADVERSE EVENTS:
Arm/Group | Insulin Lispro Protamine Suspension | Detemir
Serious Adverse Events (participants affected / at risk) | 10 | 3
Other Adverse Events (participants affected / at risk) | 93 | 86
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Insulin Lispro Protamine Suspension | Detemir
Autoimmune thyroiditis (Endocrine disorders) | 1/192 (1) | 0/189 (0)
Hyperthyroidism (Endocrine disorders) | 1/192 (1) | 0/189 (0)
Abdominal pain (Gastrointestinal disorders) | 1/192 (1) | 0/189 (0)
Mouth cyst (Gastrointestinal disorders) | 1/192 (1) | 0/189 (0)
Chest pain (General disorders) | 1/192 (1) | 0/189 (0)
Cellulitis (Infections and infestations) | 1/192 (1) | 0/189 (0)
Osteomyelitis (Infections and infestations) | 0/192 (0) | 1/189 (1)
Respiratory tract infection (Infections and infestations) | 1/192 (1) | 0/189 (0)
Diabetic foot (Metabolism and nutrition disorders) | 0/192 (0) | 1/189 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1/192 (2) | 0/189 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1/192 (1) | 1/189 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1/192 (1) | 0/189 (0)
Diabetic neuropathy (Nervous system disorders) | 0/192 (0) | 1/189 (1)
Hypoglycaemic coma (Nervous system disorders) | 1/192 (1) | 0/189 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/192 (1) | 0/189 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Insulin Lispro Protamine Suspension | Detemir
Abdominal pain upper (Gastrointestinal disorders) | 3/192 (4) | 7/189 (8)
Nausea (Gastrointestinal disorders) | 6/192 (7) | 5/189 (8)
Toothache (Gastrointestinal disorders) | 1/192 (2) | 5/189 (5)
Vomiting (Gastrointestinal disorders) | 5/192 (6) | 2/189 (2)
Fatigue (General disorders) | 2/192 (2) | 4/189 (7)
Pyrexia (General disorders) | 4/192 (5) | 0/189 (0)
Gastroenteritis (Infections and infestations) | 5/192 (5) | 3/189 (4)
Influenza (Infections and infestations) | 15/192 (16) | 16/189 (18)
Nasopharyngitis (Infections and infestations) | 27/192 (30) | 18/189 (24)
Pharyngitis (Infections and infestations) | 6/192 (6) | 4/189 (4)
Sinusitis (Infections and infestations) | 7/192 (7) | 7/189 (7)
Upper respiratory tract infection (Infections and infestations) | 0/192 (0) | 6/189 (6)
Urinary tract infection (Infections and infestations) | 3/192 (3) | 4/189 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/192 (0) | 5/189 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2/192 (3) | 4/189 (5)
Headache (Nervous system disorders) | 18/192 (32) | 14/189 (35)
Migraine (Nervous system disorders) | 5/192 (5) | 1/189 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 4/192 (16) | 3/189 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 6/192 (8) | 10/189 (12)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5/192 (5) | 5/189 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days